CLINICAL TRIAL: NCT05558124
Title: A Phase 1/1b Dose Escalation and Expansion of CPX-351 in Combination With Gemtuzumab Ozogamicin in Newly Diagnosed Acute Myeloid Leukemia
Brief Title: CPX-351 in Combination With Gemtuzumab Ozogamicin in Newly Diagnosed AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21450
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Experimental): Dose escalation to determine the maximum tolerated dose (MTD) of CPX-351 in combination with Gemtuzumab Ozogamicin in participants with newly diagnosed acute myeloid leukemia. Participants will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable. A total of 3 dose levels will be used.
  Interventions: Drug: Vyxeos; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Vyxeos — Fixed dose of Vyxeos (44 mg/m2 daunorubicin and 100 mg/m2 cytarabine) (Day 1, 3, and 5) in combination with various dose schedules of Gemtuzumab Ozogamicin (GO)
  Other Names: daunorubicin-cytarabine; CPX-351
Drug: Gemtuzumab Ozogamicin — Participants will be treated at the following dose levels:
  Dose Level 1 - Gemtuzumab Ozogamicin will administered 3mg/m2 on Day 1 Dose Level 2 - Gemtuzumab Ozogamicin will administered 3mg/m2 on Day 1 and 4 Dose Level 3 - Gemtuzumab Ozogamicin will administered 3mg/m2 on Day 1, 4, 7
  Other Names: Mylotarg

SUMMARY:
The purpose of the study is to determine the safety of combining the drugs gemtuzumab ozogamicin (GO) with CPX-351 in order to treat the disease, as well as to find the maximum tolerated dose level and recommended Phase 2 dose level of GO with a fixed dose of CPX-351.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥18 and ≤70 years with newly diagnosed any risk AML as defined by ELN 2017 criteria
* For females of child-bearing potential: use of highly effective contraception upon enrollment and during study participation and for an additional 6 months after the end of CPX-351 and Gemtuzumab ozogamicin administration: A female of child-bearing potential is considered when a sexually mature female: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months
* The effects of CPX-351 and gemtuzumab ozogamicin on the developing human fetus are unknown. For this reason, women of child-bearing potential as defined above must have a negative serum or urine pregnancy test within 24 hours prior to beginning study treatment.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* Myeloblasts expressing CD33 as determined by flow cytometry or immunohistochemistry
* ECOG ≤ 2 and eligible to receive intensive chemotherapy as determined by the treating physician
* Prior malignancy is allowed providing it does not require concurrent therapy. Exception: Active hormonal therapy is allowed.
* Prior hypomethylating agents (HMA) therapy including azacitidine or decitabine when used for non-AML diagnoses is allowed. Most recent dose must have been ≥14 days prior to day 1 of study treatment.
* Participants must have acceptable organ function
* Adequate cardiac function defined as ejection fraction of ≥50% as determined by multigated acquisition scan (MUGA) or 2D echocardiogram.
* Hydroxyurea is allowed for cytoreduction until day 1 of study treatment

Exclusion Criteria:

* Prior treatment of AML except hydroxyurea and/or leukapheresis
* Participants with acute promyelocytic leukemia (APL).
* Known current and clinically active central nervous system (CNS) leukemia.
* Severe liver disease (cirrhosis, non-alcoholic steatohepatitis, sclerosing cholangitis) or patients with known Wilson's disease.
* Participants with known active infection with hepatitis B or hepatitis C virus
* Known allergic reactions to components of the CPX-351 (cytarabine or daunorubicin) or Gemtuzumab ozogamicin.
* Patients with any prior anthracycline exposure plus any planned on-study anthracycline exposure cannot not exceed 550 mg/m2 of daunorubicin (or equivalent). For participants who have received radiation therapy to the mediastinum, the total cumulative dose of anthracycline should not exceed 400 mg/m2 of daunorubicin(or equivalent).
* Hemodynamically unstable (subjects requiring vasopressor support will not be eligible).
* Treatment with another investigational drug within 14 days.
* Uncontrolled cardiac disease including congestive heart failure class III or IV by the NYHA, unstable angina (angina symptoms at rest), new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Any disorder that compromises the subject's ability to give written informed consent and/or to comply with study procedures.
* Any substance abuse, severe and/or uncontrolled medical, social or psychiatric conditions that may prevent the subject from completing the study, interfere with the evaluation of safety and/or efficacy, or interfere with the interpretation of the study results.
* Female subject who is pregnant or breastfeeding.
* Any patient with a known FLT3 ITD or FLT3 TKD mutation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 18 Months
  Dose escalation will determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Vyxeos plus Gemtuzumab Ozogamicin. The MTD is the highest dose of the combination therapy that dose not cause unacceptable side effects.

SECONDARY OUTCOMES:
Rate of Complete Remission | Up to 18 Months
  Rate of complete remission (CR) and complete remission with incomplete blood count recovery (CRi). The definition of CR and CRi is based on the European LeukemiaNet 2017 Response Criteria for AML.
Measurable Residual Disease | Up to 18 Months
  Rate of measurable residual disease via RT-PCR for core binding factor leukemia as well as NPM1 mutated AML
Overall Survival | Up to 5 years
  Overall survival is defined as the duration of time from start of treatment to the time of death from any cause or date of last contact.
Relapse Free Survival (RFS) | Up to 18 Months
  RFS is defined as time interval between achievement of CR to time of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Onyee Chan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE